CLINICAL TRIAL: NCT04603573
Title: Clinical and Cost-effectiveness of Fluoride Varnish Versus Resin Based Fissure Sealant in Newly Erupted Permanent Molars in Group of Egyptian Children : A Randomized Clinical Trial ( Part 1)
Brief Title: Clinical and Cost-effectiveness of Fluoride Varnish Versus Resin Based Sealant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Zaghloul, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112
Record Dates: First submitted 2020-10-13; First posted 2020-10-27 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-01

CONDITIONS: Cost Effectiveness

STUDY DESIGN:
Intervention Model Description: The study will be randomized, allocation-blinded, two-arm, parallel-group trial. The participants will be randomized on a 1: 1 allocation ratio to receive one of the following interventions:
  * Resin-based fissure sealant FS.
  * Fluoride varnish FV
Masking Description: No one is blinded ( unfortunately) as fissure sealant will be obvious
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (intervention) (Experimental): Fluoride varnish (3M Clinpro White Varnish 5% sodium fluoride). Group (1)
  Interventions: Device: fluoride varnish (3M Clinpro White Varnish 5% sodium fluoride )
- comparator (Active Comparator): Resin based fissure sealant (3M Clinpro Sealant, light cure, low viscosity, fluoride release).group (2)
  Interventions: Device: Resin based fissure sealant (3M Clinpro sealant )

INTERVENTIONS:
Device: fluoride varnish (3M Clinpro White Varnish 5% sodium fluoride ) — 5% Sodium Fluoride Varnish is a fluoride varnish which is applied to tooth surfaces for sealing dentinal tubules and treatment of hypersensitive teeth. The varnish is applied in a thin layer over the tooth with an applicator brush, and moisture from saliva cures the varnish for adhesion to the tooth surface.
  Other Names: 5% Sodium Fluoride Varnish 3M
  Arms: (intervention)
Device: Resin based fissure sealant (3M Clinpro sealant ) — teeth will be isolated with coton rolls and saliva ejector then etching for pits and fissure then tooth will be washed then apply resin based fissure sealant on occlusal surface.
  resin fissure sealant is a more sensitive for saliva.
  Other Names: resin fissure sealant 3M
  Arms: comparator

SUMMARY:
The aim of the present study is determine the cost-effectiveness, clinical-effectiveness, acceptability and adverse effect of resin sealants versus the fluoride varnish for the prevention of dental caries on newly erupted permanent molars.

DETAILED DESCRIPTION:
A Cochrane systematic reviews found low quality evidence supporting Current practice guidelines that recommend the use of Resin based fissure sealant over Fluoride varnish in prevent dental caries. However, they did not address the cost-effectiveness, A more recent systematic review and meta-analysis concluded that no statistical significance difference between Resin based fissure sealant and Fluoride varnish with a high-quality evidence in prevent dental caries.

This trial will measure cost effectiveness and clinical effectiveness for resin fissure sealant and fluoride varnish.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children with no physical or mental disorders. Children with newly fully erupted permanent molars (PMs).

Exclusion Criteria:

* Teeth will be excluded from the study if they had any of the following:

  * Dental caries in dentine
  * History of pain or swelling. Parents refused their children participate in the trial

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Clinical-effectiveness (will be measured with DFS | Through study completion, an average of one year
  Clinical-effectiveness (will be measured by DFS) Clinical effectiveness (continuous outcome will be measured with DFS D Decayed in permanent molar Filling in permanent molar S Surface

SECONDARY OUTCOMES:
Cost-effectiveness (will be measured with Incremental cost effective ratio ICER | through study completion, an average of one year
  Cost-effectiveness (will be measured with Cost-effectiveness will be calculated based on the following measures:-
  Economic measures (continuous outcome, (money) will be measured with Calculate The total cost of each of FV and FS in every visit) .
  Clinical effectiveness (continuous outcome will be measured with DFS.
Time of application (continuous outcome, (minutes) will be measured with stopwatch. | Through application of interventions in treatment visit( baseline)
  Time of application (continuous outcome, (minutes) will be measured with stopwatch.
acceptability will be measured by questionnaire | through study completion, an average of one year
  I will ask the parent and child if this trial is acceptable or not
adverse effect will be measured by questionnaire | through study completion, an average of one year
  Questionnaire for the parent (allergy, diarrhea or vomiting )

CONTACTS AND LOCATIONS:
Locations (1):
- Oral and dental medicine Cairo university, Giza, Egypt